CLINICAL TRIAL: NCT04443283
Title: A Prospective Cohort Study on the Effect of Latent Infection of Tuberculosis on the Pregnancy Outcome of IVF-ET in Infertile Patients With Radiographic Lesions Suggesting Old Healed Tuberculosis
Brief Title: The Effect of Latent Tuberculosis Infection on the Pregnancy Outcome of IVF-ET
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PCCMRP
Record Dates: First submitted 2020-06-21; First posted 2020-06-23 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-03

CONDITIONS: Infertility; Tuberculosis
Keywords: infertility; IVF-ET; old tuberculosis; pregnancy outcome; latent tuberculosis infection
MeSH Terms: conditions — Infertility; Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — collect seum sample to detect some inflammatory factors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LTBI Group: IGRA(+)
  Interventions: Other: No intervention
- No LTBI Group: IGRA(+)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a observation study, with no intervention

SUMMARY:
This study evaluate the effect of latent infection of tuberculosis on the pregnancy outcome of IVF-ET in infertile patients with radiographic lesions suggesting old healed tuberculosis

DETAILED DESCRIPTION:
China is one of the countries with high burden of tuberculosis (TB) defined by WHO. IVF-ET is an effective method to treat infertility. Chest X-ray is a routine examination before IVF-ET, which can exclude active tuberculosis. However, for patients with chest X-ray showing old healed tuberculosis, the relationship between latent tuberculosis infection (LTBI) and pregnancy outcomes is unknown. In this study, a prospective cohort study was carried out in infertile women who were planning to receive IVF-ET. IGRA were tested in patients with old tuberculosis in chest X-ray. A cohort of IGRA positive and IGRA negative was constructed. The pregnancy outcomes were followed up prospectively and the relationship between latent infection of tuberculosis and pregnancy outcomes was analyzed. The primary outcome was clinical pregnancy rate, miscarriage rate and live birth rate. Secondary outcomes were tuberculosis reactivation during pregnancy period and in 3 months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* The patients who referred to the reproductive center for IVF-ET
* Chest radiography showed old healed tuberculosis

Exclusion Criteria:

* active tuberculosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were recruited between January 1, 2019, and December 30, 2020, at Peking University Third Hospital, a tertiary referral hospital in Beijing, China. A board-certified radiologist reviewed CXRs and, if available, chest computed tomography (CT) scans, of women who referred to the reproductive center for IVF-ET. The patients who had chest imaging abnormalities consistent with old healed TB were admitted or referred to the respiratory clinic and enrolled.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 30 days after the ET procedure
  Clinical pregnancy was defined as the observation of a gestational sac on ultrasonography. The clinical pregnancy rate was defined as clinical pregnancy per embryo transfer.
miscarriage rate | 40 weeks after the ET procedure
  Miscarriage was defined as a pregnancy loss before 28 weeks of gestation (calculated among women who became pregnant). The miscarriage rate was defined as miscarriages per clinical pregnancy.
live birth rate | 40 weeks after the ET procedure
  Live birth was defined as delivery of a living foetus (or living foetuses) beyond 28 weeks of gestation. The live birth rate was defined as live birth per embryo transfer.

SECONDARY OUTCOMES:
tuberculosis reactivation | 40 weeks after the ET procedure
  tuberculosis during pregnancy period and in 3 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ji Qiao, MD., Principal Investigator — Reproductive Medicine Centre，Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gai X, Chi H, Zeng L, Cao W, Chen L, Zhang C, Li R, Sun Y, Qiao J. Impact of Positive Interferon-Gamma Release Assay on IVF-ET Pregnancy Outcomes in Infertile Patients With Untreated Prior Tuberculosis: A Prospective Cohort Study. Front Med (Lausanne). 2021 Nov 16;8:749410. doi: 10.3389/fmed.2021.749410. eCollection 2021. PMID 34869442